CLINICAL TRIAL: NCT03990415
Title: Physical Function in Older Adults in the Stay Strong, Stay Healthy Program
Brief Title: Stay Strong, Stay Healthy Outcomes in Older Adults
Acronym: MU-SSSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana Duren (Other)
Responsible Party: Sponsor-Investigator, Dana Duren, Professor and Director of Orthopaedic Research at the Missouri Orthopaedic Institute, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014256
Record Dates: First submitted 2019-06-06; First posted 2019-06-19 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Frail Elderly; Sedentary Lifestyle
Keywords: Elderly; Balance; Strength Training
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into three groups of equal size. The experimental group (Stay Strong, Stay Healthy strength training program), the walking exercise group, and the sedentary control group will participate in the trial in parallel for up to ten weeks. After the intervention period, participants from each group will have the opportunity to participate in an interview about their experiences.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator (Dr. Duren) will randomize participants into each of the three study groups. The research team responsible for assessments and analysis will be blinded to each participant's assignment. Dr. Duren will unblind the research team after the intervention period and data collection and analysis has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stay Strong, Stay Healthy Group (Experimental): The Stay Strong, Stay Healthy strength training group will meet two times per week for an hour, for eight consecutive weeks. This class provides participants a structured program to learn and progress through strength training exercises designed to increase overall fitness, flexibility, and balance.
  Interventions: Behavioral: Exercise
- Walking Group (Active Comparator): The walking group will meet two times per week for an hour, for eight consecutive weeks. This class provides participants a structured walking program to help delineate the effects of the strength training program and exercise in general.
  Interventions: Behavioral: Exercise
- Delayed Start Group (No Intervention): The delayed start group will not make any changes to their sedentary lifestyle and will be encouraged to not begin any exercise programs throughout the duration of the study.

INTERVENTIONS:
Behavioral: Exercise — Exercise is a behavioral intervention, the primary aim of this investigation is to elucidate if strength training is a more effective exercise intervention than walking for the improvement of balance in older adults.
  Arms: Stay Strong, Stay Healthy Group; Walking Group

SUMMARY:
The University of Missouri's Stay Strong, Stay Healthy (SSSH) program is an eight week strength training class for older adults. Exercise training programs, like SSSH, can increase muscle mass and strength, improve bone density and reduce the risk of osteoporosis and related fractures, improve diabetes, heart disease, arthritis, depression, and obesity; and increase self-confidence, sleep and vitality in older adults. Specifically, the SSSH program has been shown to increase elderly individuals' confidence in their physical abilities. The primary objective of this research study is to track physiologic changes and determine the effectiveness of the SSSH exercise intervention to improve balance and fall risk in older adults. Participant's balance, gait, muscle strength, body composition, and skeletal health will be compared to a walking group and to a sedentary control group prior to and immediately following the eight week exercise intervention. After the intervention period participants will have the opportunity to participate in an interview process to further discuss their experiences and perceptions regarding the intervention and their health.

DETAILED DESCRIPTION:
Research Background and Objectives The University of Missouri's Stay Strong, Stay Healthy (SSSH) program is an eight week strength training class for older adults. SSSH is modeled after the evidence-based StrongWomen program developed by researchers at Friedman School of Nutrition Sciences at Tufts University. While the original Tufts program included only women, University of Missouri Extension has adapted the curriculum to also include men. Strength training programs, like SSSH, can increase muscle mass and strength, improve bone density and reduce the risk of osteoporosis and related fractures, improve diabetes, heart disease, arthritis, depression, and obesity; and increase self-confidence, sleep and vitality in older adults. Specifically, the SSSH program increases elderly individuals' confidence in their physical strength and balance. The present study will elucidate the effects of the SSSH program on specific measures of balance, muscle capacity, and skeletal health in a cohort of older adults from Central Missouri.

The primary objective of the quantitative part of the research study is to track physiologic changes and determine the effectiveness of the SSSH exercise intervention in older adults. Participant's balance, gait, muscle strength, body composition, and skeletal health will be compared to a walking group and to a sedentary control group prior to and immediately following the eight week exercise intervention.

Participant centered objectives include:

* Participants will improve their balance, thus reducing their risk for falls.
* Participants will increase their muscle strength and improve body composition.
* Participants will increase their rate of bone formation.
* Participants will improve their cognition and sleep habits.
* Participants will increase their physical activity

The primary objective of the qualitative part of the research study is to explore perceptions of the impact of physical activity and changes in behaviors and attitudes of participants who completed the intervention period. The sequential approach of this study will (1) explore the effects of participating in the Stay Strong, Stay Healthy study that were difficult to measure quantitatively and (2) help interpret the quantitative findings and understanding.

Topics that will guide the qualitative study include participants':

* Concerns, motivations/benefits, and needs/barriers to physical activity
* Perceptions of social influences on physical activity
* Perceptions of impact of physical activity on psychological and emotional well-being, cognition, and sleep
* Perceptions of confidence related to fear of falling
* Perceptions of changes in behaviors and attitudes based on bone density test results

Recruitment Process The Stay Strong, Stay Healthy program is conducted throughout the state of Missouri. Class sessions are advertised by posting flyers and in newspapers. At the University of Missouri-Columbia, the SSSH program is advertised by posting flyers around campus and utilizing the email group for retired MU employees. Dr. Baker and research staff will also present the research study participation opportunity at pre SSSH sessions in Columbia and surrounding areas. The investigators will be available to answer questions via email and phone for any potential participants prior to their first visit on campus. The inclusion and exclusion criteria listed below in addition to the PAR-Q form will make up the initial screening form. During the recruitment process research staff will use this form to quickly screen potential participants for overt exclusion criteria, thus reducing the number of "screen failure" participants who will have to coordinate travel to campus for the first consenting visit. No personal health information is contained in these forms and all questions are yes/no, and this data will only be recorded for screening failures to inform selection bias. The inclusion of this form is purely the research team's attempt to reduce patient burden as travel can be very difficult for this patient population.

Consent Process Only research staff cleared to obtain written consent will escort participants to a private room in Gwynn Hall, where all screening and consenting will take place. After participants have cleared the initial screening checklist (the PAR-Q form and inclusion/exclusion criteria), research staff will deliberately and clearly explain each aspect of the informed consent. Participants will be encouraged to ask questions and will be reminded of the voluntary nature of their participation prior to signing the informed consent form. Signed informed consents will be collected and securely stored in Dr. Duren's office. At this time, participants will also be given an additional copy of the informed consent for future reference. At the end of the intervention participants will be reconsented to participate in the interview process if they choose.

Number of Subjects Using G*Power (V3.1) sample size calculations were completed using estimated and calculated effect sizes from previously published SSSH research 7-9. Estimated low and medium effect sizes resulted in a sample size ranging from 12-55. Calculated effect sizes for the 30 second sit to stand (balance), DXA (body composition), and the Self Administered Gerocognitive Examination (cognitive function) resulted in a sample size ranging from 9 to 43. The investigators believe nearly 50 participants total are needed to reach statistical power for this study; however, assuming 15% attrition rates, 60 participants (up to 20 per group) will be recruited for the study.

Study Procedures/Design/Treatment Plan Participants who chose to enroll will be required to provide approximately five hours minimum or up to seven hours maximum of their time total, in addition to intervention exercise activities. The first visit will consist of the initial screening form and the informed consent, followed by a facility tour, and familiarization of the testing procedures and will take one hour. The second and third visits are identical in procedure and time required and will consist of a urine sample, blood draw, anthropometrics, DXA scans, and functional performance assessments, and questionnaires. These two visits lasting 2 hours each will occur immediately before and after the eight week intervention period. The last potential visit will be for follow-up interviews. Each visit and all questionnaires and procedures are explained in greater detail below.

Potential Risks/Adverse Events

The research team has taken extensive measures to reduce risk and the potential for adverse events. Both participant and research staff safety are a priority. The investigators will minimize these risk by taking the following precautions:

* Standard aseptic technique will be used for drawing blood and only trained personnel will complete blood sample, DXA scans, and functional testing.
* This research does not involve vulnerable populations and the investigators are not collecting any highly sensitive personal or medical information (e.g. social security numbers, banking information, HIPAA information) and do not expect any of the collected data to impact a participant's employment, insurability, social status, or reputation if it were to become public.
* Subjects' information will be coded and will be stored on University of Missouri secure database and the investigators will follow a strict protocol to ensure patient confidentiality at all times.
* Subjects are asked to perform balance assessment tests close to a wall under the supervision of trained personnel to avoid falls. Trained research staff will always be within reach to aid a participant if they lose their balance. Participants will never be left alone to complete a task.

During follow-up interviews, audio recording will be used for data collection. We will request that participants not identify anyone during their interview and the transcriptions of the audio recordings will be de-identified if participants do not heed our request. During the interview, participants may become tired from answering questions and talking or become frustrated by difficulty communicating as you want. The interviewer will listen to the participant closely and carefully and ask him/her to let her know if they become uncomfortable during the study and offer the participant breaks, as needed.

Any serious adverse events will be reported directly to the IRB, please see the Data Safety Monitoring Plan below for more details. In case of emergency, the electromyography, dual x-ray absorptiometry, or blood drawing process will be immediately stopped. The investigators will dial 911 in the case of emergency.

Anticipated Benefits Potential benefits experienced by the participant include: decreased risk of fall and frailty; improve sleep and cognition; increased muscle mass and strength; and improvements in bone turnover rates. Potential benefits to society include the curbing of the declining physical and mental capacity among seniors, which are key risk factors for falls. Strength training has been shown to mitigate these factors in seniors, ultimately saving the healthcare system billions of dollars in associated costs. Participants may gain a sense of accomplishment for helping us better understand the impact of the Stay Strong, Stay Healthy program.

Costs The costs for this study and procedures will be paid through internal departmental grant funding through the Department of Nutrition and Exercise Physiology, University of Missouri-Extension, and the Missouri Orthopaedic Institute.

Data Safety Monitoring Plan In order to protect the participants' personal information, data, and right to privacy this research team will take extensive precautions to maintain confidentiality. After the participant has cleared the initial screening forms and signed the informed consent all remaining surveys, questionnaires, DXA results, blood samples, and data sheets will only contain the participant' identification code. The key linking names and participant identification codes will be accessible to Dr. Dana Duren and she will only share the key with the research team once unblinding is necessary. All paper records will be kept in a locked filing cabinet in Dr. Duren's MU office (she is a Professor and Director of Orthopaedic Research and is familiar with handling confidential documents). Computerized records of experimental data will be similarly coded and will be maintained on a password protected MU secure computer. Copies of signed consent forms, as well as the experimental log book, are kept in a locked file cabinet in Dr. Duren's office. Participants will not be individually identified in any publications.

Additionally, all adverse events and/or unanticipated problems will be evaluated by Drs. Duren, Ball, and Baker as they occur, for subject safety and appropriate follow-up assessment, treatment, or care. All adverse events and/or unanticipated problems will be evaluated and assessed to answer the following questions: Is the event unexpected? Is the event related or possibly related to participation in the research? Does the event suggest that the research places subjects or others at a greater risk of harm than previously known or recognized? If all three answers are "yes", the event will be reported to the IRB within 5 days of the investigator becoming aware of the event. While reviewing each event, the PI(s) will determine if it is safe for the subject to continue participating in the trial and if it is safe to continue enrollment and research activity for all subjects.

Multiple Sites University of Missouri is the only site where research activities will occur. All required approvals are in order for the three specific rooms where data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female ≥60 years of age
* Are sedentary (no strength training and <30min/wk of other physical activity in the past 3 months)
* Are ambulatory (cane or walker permitted)
* Are free from current physical injury or illness preventing physical activity

Exclusion Criteria:

* Answered YES to two or more questions on the PAR-Q form
* Are female subjects who have not fully gone through menopause
* Were a previous SSSH participant
* Have dementia/Alzheimer's or other cognitive impairments that would limit ability to follow directions

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana L Duren, PhD, Principal Investigator — Director of Orthopaedic Research at the University of Missouri
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seguin RA, Economos CD, Hyatt R, Palombo R, Reed PN, Nelson ME. Design and national dissemination of the StrongWomen Community Strength Training Program. Prev Chronic Dis. 2008 Jan;5(1):A25. Epub 2007 Dec 15. PMID 18082014
- [Background] Seguin RA, Folta SC, Nelson ME, Hanson KL, LaCroix AZ. Long-Term Body Weight Maintenance among StrongWomen-Healthy Hearts Program Participants. J Environ Public Health. 2017;2017:4372048. doi: 10.1155/2017/4372048. Epub 2017 Mar 2. PMID 28352287
- [Background] Guizelini PC, de Aguiar RA, Denadai BS, Caputo F, Greco CC. Effect of resistance training on muscle strength and rate of force development in healthy older adults: A systematic review and meta-analysis. Exp Gerontol. 2018 Feb;102:51-58. doi: 10.1016/j.exger.2017.11.020. Epub 2017 Nov 28. PMID 29196141
- [Background] Foster C, Armstrong MEG. What types of physical activities are effective in developing muscle and bone strength and balance? J Frailty Sarcopenia Falls. 2018 Jun 1;3(2):58-65. doi: 10.22540/JFSF-03-058. eCollection 2018 Jun. PMID 32300694
- [Background] Beavers KM, Walkup MP, Weaver AA, Lenchik L, Kritchevsky SB, Nicklas BJ, Ambrosius WT, Stitzel JD, Register TC, Shapses SA, Marsh AP, Rejeski WJ. Effect of Exercise Modality During Weight Loss on Bone Health in Older Adults With Obesity and Cardiovascular Disease or Metabolic Syndrome: A Randomized Controlled Trial. J Bone Miner Res. 2018 Dec;33(12):2140-2149. doi: 10.1002/jbmr.3555. Epub 2018 Aug 7. PMID 30088288
- [Background] Northey JM, Cherbuin N, Pumpa KL, Smee DJ, Rattray B. Exercise interventions for cognitive function in adults older than 50: a systematic review with meta-analysis. Br J Sports Med. 2018 Feb;52(3):154-160. doi: 10.1136/bjsports-2016-096587. Epub 2017 Apr 24. PMID 28438770
- [Background] Syed-Abdul, M.M., Peterson, E.C., Mills-Gray, S.L., Parks, E.J. & Ball, S.D. Stay Strong, Stay Healthy: University of Missouri-Extension's Strength-Training Program for Older Adults in Community Settings. Med Sci Sports Exer 48:5, 125-125 (2016).
- [Background] Crowe EM, Ball SD. Effectiveness of Advanced Stay Strong, Stay Healthy in Community Settings. Gerontol Geriatr Med. 2015 Aug 3;1:2333721415596462. doi: 10.1177/2333721415596462. eCollection 2015 Jan-Dec. PMID 28138461
- [Background] Ball S, Gammon R, Kelly PJ, Cheng AL, Chertoff K, Kaume L, Abreu EL, Brotto M. Outcomes of Stay Strong, Stay Healthy in community settings. J Aging Health. 2013 Dec;25(8):1388-97. doi: 10.1177/0898264313507318. Epub 2013 Oct 22. PMID 24150062
- [Derived] Baker BS, Weitzel KJ, Royse LA, Miller K, Guess TM, Ball SD, Duren DL. Efficacy of an 8-Week Resistance Training Program in Older Adults: A Randomized Controlled Trial. J Aging Phys Act. 2021 Feb 1;29(1):121-129. doi: 10.1123/japa.2020-0078. Epub 2020 Aug 12. PMID 32788412
- See also: The home SSSH link — https://extension2.missouri.edu/programs/stay-strong-stay-healthy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study team aimed to recruit 60 participants (20 per study arm) that met all eligibility criteria. Participants were recruited from the local University, churches, assisted living facilities, and the senior center. Recruitment efforts began in late May, 2019 and ended in late June, 2019.
Period: Overall Study
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Started | 19 | 19 | 14
Completed | 15 | 17 | 14
Not Completed | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 20 participants were recruited in each group. Before study arm assignment a single SSSH participant was excluded for being too active and a single Walk participant was excluded due to cognitive impairment. After study arm assignment three participants from the delayed start group dropped out once they were assigned their group, one due to cognitive impairment, one due to general voluntary termination, and one due to an unexpected surgical procedure unrelated to study participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group | Total
Number analyzed (Participants) | 19 | 19 | 14 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (8.0) | 69.4 (9.2) | 67.6 (7.0) | 68.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 10 | 39
  Male | 5 | 4 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 19 | 19 | 14 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 14 | 52
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.1 (6.1) | 30.5 (7.5) | 31.2 (8.4) | 32.0 (7.4)
Minutes per week of Physical Activity [Mean (Standard Deviation); unit: minutes per week] | 41.8 (49.7) | 42.2 (55.0) | 65.0 (55.7) | 48.2 (53.3)
Number of falls in the past year [Mean (Standard Deviation); unit: falls per year] | 1.0 (1.9) | 0.6 (0.9) | 2.0 (2.4) | 1.1 (1.8)
Fear of falling score [Mean (Standard Deviation); unit: units on a scale] — The fear of falling score ranges from 1-4, with 1 being no fear and 4 being the most fear.
  units on a scale | 2.2 (1.0) | 2.1 (0.7) | 2.0 (1.0) | 2.1 (0.9)
Sleep Quality [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index is a survey ranging from 0-21. Higher scores are worse and scores under 5 indicate good sleep.
  units on a scale | 5.6 (2.7) | 5.8 (3.3) | 5.9 (3.0) | 5.7 (3.0)
Cognition Scores [Mean (Standard Deviation); unit: units on a scale] — The SGE cognition test ranges from 0-21. Scores above 17 are considered normal.
  units on a scale | 18.3 (2.2) | 18.0 (2.5) | 18.6 (2.2) | 18.3 (2.3)
30STS reps [Mean (Standard Deviation); unit: repetitions] — The 30 second sit-to-stand measures the number of full repetitions the participant can stand fully from a chair and then sit down again in 30 seconds. High numbers indicate greater fitness and leg strength.
  repetitions | 9.1 (4.5) | 8.9 (2.6) | 9.2 (3.5) | 9.1 (3.6)
TUG time in seconds [Mean (Standard Deviation); unit: seconds] — The timed-up-and-go measures the time it takes to go from a seated position to standing, then walk around a marker 8 feet away, and return to the seated position. Longer times are indicators or slower gait speed, worse balance/coordination, and reduced lower body strength.
  seconds | 9.9 (5.0) | 8.5 (2.3) | 9.5 (3.9) | 9.3 (3.9)
10 meter walk test [Mean (Standard Deviation); unit: seconds] | 6.9 (2.4) | 6.1 (1.0) | 6.6 (2.2) | 6.5 (2.0)
Grip Strength (mean) [Mean (Standard Deviation); unit: kg] — Mean grip strength is the average amount of force in kg that each hand was able to produce - called grip strength.
  kg | 28.9 (9.5) | 26.5 (8.5) | 28.3 (12.0) | 27.8 (9.8)
Mean Back-Scratch Flexibility [Mean (Standard Deviation); unit: inches] — Mean back-scratch is a test of upper body flexibility. The higher the average score the more flexible, if the score is low or negative that indicates less or poor upper body flexibility.
  inches | -6 (4.5) | -5.3 (5.6) | -7.5 (5.2) | -6.2 (5.1)
Mean Sit-n-reach Flexibility [Mean (Standard Deviation); unit: inches] — Mean sit-n-reach is a test of lower body flexibility. The higher the average score the more flexible, if the score is low or negative that indicates less or poor lower body flexibility.
  inches | 1.7 (4.3) | -1.4 (5.2) | -2.6 (5.1) | -.6 (5.1)
Mean CDC 4 static balance test [Mean (Standard Deviation); unit: seconds] — The CDC balance test has individuals complete four stances for up to 10 seconds. If a participant can only maintain the stance without help for less than 10 seconds it may indicate balance impairments and an increased risk of falling. Scores of 40 are ideal as that means they completed all four stances for the full 10 seconds.
  seconds | 31.6 (7.6) | 33.7 (6.8) | 34.3 (7.6) | 33.1 (7.3)
Bone Mineral Density T- Score [Mean (Standard Deviation); unit: T-Score] — Bone mineral density is how we calculate is a person has the clinical diagnosis of osteopenia or osteoporosis. Lower and negative numbers indicate less bone mass while positive and larger numbers indicate greater bone mass compared to reference population. For T-Scores scores above -1.0 indicate normal bone mass and scores under -2.5 indicate osteoporosis.
  T-Score | -1.2 (0.9) | -1.9 (1.6) | -1.8 (1.7) | -1.6 (1.4)
Bone Turnover Marker Ratio [Mean (Standard Deviation); unit: Ratio] — This is the ratio of PINP and CTX. PINP indicates bone formation and CTX indicates bone resorption. Larger numbers indicate more positive bone growth and smaller numbers indicate more bone is being resorbed.
  Ratio | 40.3 (22.9) | 43.7 (22.3) | 49.9 (22.9) | 44.3 (23.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance During a Dynamic Task Using Force Plates.
Description: Participants will complete the 30 second sit-to-stand dynamic balance task on two force plates, which will allow for a sensitive measure of balance. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Population: One delayed start participant did not complete the post task due to knee pain.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 13
percentage of change | 32.4 (24.8) | 18.1 (24.6) | 10 (25.1)

2. Primary Outcome: Change in Balance During a Static Task Using Force Plates.
Description: Participants will complete the CDC 4 stance static balance task on force plates, allowing for a more sensitive measure of balance. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | 3.3 (29.1) | 9.3 (29.1) | 5.4 (28.1)

3. Secondary Outcome: Changes in Grip Strength Using a Hand Dynamometer.
Description: Participants will test their grip strength using a hand dynamometer over time. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | -1.3 (29.4) | -9.8 (34.5) | 0.3 (11.6)

4. Secondary Outcome: Changes in Walking Speed Using a 10 Meter Course.
Description: Participants will walk a self selected pace over a 10 meter distance and the investigators will time this process before and after the intervention. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | -6.1 (6.8) | -5.5 (7.3) | -1.2 (7.4)

5. Secondary Outcome: Changes in the Timed Up and Go
Description: Investigators will test the change in participant's timed up and go (TUG) performance. This is the TUG that covers an 8 foot distance. The pre and post measure will be used to calculate a percent change, with positive values indicating a decline in performance and a negative value indicating an improvement in performance times.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | -8.1 (10.6) | -8.5 (10.9) | -6.5 (11.0)

6. Secondary Outcome: Changes in Upper Body Muscle Flexibility Using the Back Scratch Test.
Description: Investigators will test the change in participant's upper body flexibility by using the back scratch test. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Population: One delayed start participant did not complete the post testing due to shoulder pain.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 13
percentage of change | -105.2 (38.5) | -13.6 (41.1) | 11.7 (41.0)

7. Secondary Outcome: Changes in Lower Body Muscle Flexibility Using the Sit and Reach Test.
Description: Investigators will test the change in participant's lower body flexibility by using the sit and reach test. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | 59.7 (196.7) | 108.5 (221.5) | 13.5 (175.6)

8. Secondary Outcome: Changes in Sleep Quality Using the Pittsburgh Sleep Quality Index Test.
Description: Participants will complete the Pittsburgh Sleep Quality Index Test. The pre and post measure will be used to calculate a percent change, with positive values indicating an increase and a negative value indicating a decline which is good.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | -19.9 (49.2) | 17.2 (37.7) | 54.6 (38.3)

9. Secondary Outcome: Changes in Cognition Performance Using the Self Administered Gerocognitive Examination.
Description: Participants will complete the Self Administered Gerocognitive Examination. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 14
percentage of change | -0.9 (57.6) | 0.3 (42.8) | 0.2 (39.8)

10. Secondary Outcome: Changes in Bone Activity Using the Ratio of Serum Bone Turnover Markers (PINP ng/mL and CTX ng/mL).
Description: We will test the change in bone activity by using blood samples to measure markers of bone formation (PINP) and bone resorption (CTX). The percent change in the ratio will allow us to see the extent of bone resorption occurring with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Population: We were not able to retrieve a blood sample from one delayed start participant.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 15 | 17 | 13
percentage of change | 268.3 (75.8) | 25.2 (78.6) | 61.8 (92.4)

11. Secondary Outcome: Changes is Bone Mineral Density T-scores
Description: aBMD measures of bone mineral density and their associated t-scores from the DXA. The pre and post measure will be used to calculate a percent change, with positive values indicating an improvement and a negative value indicating a decline.
Time Frame: Baseline and at end of intervention period, typically 8 weeks.
Population: Individuals who have metal implants did not have this calculation completed.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
Number analyzed (Participants) | 11 | 13 | 10
percentage of change | -127.3 (23.2) | -152.9 (26.4) | -138.5 (24.8)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Same definition
Arm/Group | Stay Strong, Stay Healthy Group | Walking Group | Delayed Start Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03990415/Prot_SAP_000.pdf